CLINICAL TRIAL: NCT04993989
Title: Pharmacy-based Study on the Effectiveness, Tolerability, Usage Behavior and User Satisfaction of Iberogast® in Functional and Motility-related Gastrointestinal Diseases, Preferably Irritable Bowel Syndrome.
Brief Title: A Pharmacy-based Study to Learn More About How Well Iberogast Works, How it Affects the Body, How it is Used, and User Satisfaction in Patients With Functional and Motility-related (Stomach and Bowel Movement-related) Gastrointestinal Diseases, Including Irritable Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21971
Record Dates: First submitted 2021-06-30; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Functional and Motility Related Gastrointestinal Disorders Such as Irritable Bowel Syndrome and Functional Dyspepsia
Keywords: Iberogast; Functional dyspepsia; Irritable bowel syndrome; Stomach mucosal inflammation; Pharmacy based survey
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — iberogast

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pharmacy based survey: Patients received a questionnaire, which was filled out and returned to the Contract Research Organization (CRO) or, alternatively to the pharmacy.
  Interventions: Drug: Iberogast (STW5, BAY98-7411)

INTERVENTIONS:
Drug: Iberogast (STW5, BAY98-7411) — Survey without any intervention assigned in the study.

SUMMARY:
Researchers want to learn more about the day-to-day use of Iberogast in people who have functional and motility-related gastrointestinal (stomach and bowel) diseases.

Functional and motility-related stomach and bowel diseases are conditions in which the functionality of the gut, mainly the gut muscles or the gut/brain axis is disturbed. Functional and motility related stomach and bowel diseases cause symptoms like heartburn, cramps and u pain of the upper and middle part of the belly, also known as functional dyspepsia (FD), and irritable bowel syndrome (IBS). IBS affects predominantly the lower digestive system and causes symptoms like pain of the belly, cramps, bloating, diarrhea, and constipation.

In this study, the researchers want to learn more about Iberogast, a plant-based treatment. Iberogast is available to treat stomach and bowel diseases such as FD and IBS.

Earlier studies with Iberogast have shown how well it works and how it affects the body. But, little is known about the day-to-day use of Iberogast and how satisfied patients are who take it. So in this study, the researchers want to learn more about Iberogast including:

* how well it works in day-to-day use
* how it affects the body, also referred to as tolerability
* how it is used day-to-day
* how safe it is
* how satisfied patients are who take it

To answer these questions, the researchers will collect information from pharmacies in Germany. Patients who get Iberogast from these pharmacies to help treat their gastrointestinal disease will complete a questionnaire before, during and after taking Iberogast. The researchers will use the results from the questionnaires to learn more about:

* the disease details of the patients who are taking Iberogast
* the patients' symptoms while taking Iberogast
* if the patients' symptoms change after taking Iberogast
* how satisfied patients are with Iberogast
* if the patients had adverse events

An adverse event is any medical problem that a participant has during a study.

This study will include patients in Germany who:

* have functional stomach and bowel symptoms or disorders like FD or IBS
* take Iberogast to treat symptoms of their stomach and bowel disease
* are able to complete the questionnaire

There will be no required tests or visits with a study doctor in this study. No treatments will be given as part of this study. The researchers will review information collected from patients who have decided for their own or by recommendation of their doctors or pharmacist to take Iberogast. The researchers will collect the results from the patient questionnaires from November 2017 to March 2018.

ELIGIBILITY:
Inclusion Criteria:

* Patients received a questionnaire, if all of the following applied:

  * Patients intent to use Iberogast® for the treatment of functional gastrointestinal symptoms (e.g. stomach pain, abdominal cramps, nausea, bloating, flatulence and heartburn) as well as defined functional dyspepsia (FD) and irritable bowel syndrome (IBS).
  * Patients suffered more from intestine-related complaints
  * Patients expressed their interest in participating in the study
  * Patients were willing and able to answer the questionnaire completely and plausibly

Exclusion Criteria:

* Patients did not receive a questionnaire, if

  * Patients did not currently use Iberogast® to treat gastrointestinal diseases such as irritable stomach and irritable bowel syndrome (medicine cabinet & travel medicine cabinet) or bought the product for someone else
  * Patients did not give a specific reason for treatment
  * Patients did not show interest in participating
  * Patients suffered exclusively from diarrhea and constipation
  * Patients suffered exclusively from heartburn.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: German patients who used Iberogast for treatment of gastrointestinal complaints.
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Onset of symptom improvement as assessed by patients | At baseline
  Patients answered how quickly a significant improvement in their gastrointestinal symptoms was felt after taking Iberogast.
Symptom improvement as assessed by patients. | 7 days
  Patients assessed the improvement in symptoms/concomitant complaints on an 5 -point Likert scale from 0=no improvement, 1=mild improvement, 2=moderate improvement, 3=good improvement, to 4=very good improvement.
Effectiveness of Iberogast in comparison to other treatments as assessed by patient. | 7 days
  Patients indicated the respective medication they used/ consumed earlier for their complaints on an 3 -point rating scale as "better", "same" and "poorer".
Number of participants with gastrointestinal complaints ,categorized by severity. | 7 days
  Patients assessed tolerability with Iberogast on 5-point Likert scale as "very good", "good", "medium", "poor", and "very poor''.
Patients´ usage behavior as assessed by patients. | At baseline
  Patients answered why Iberogast was chosen and what was the source of awareness of the product.
Number of participants with adverse events. | 7 days
Patients 'satisfaction as assessed by patients. | 7 days
  Patients assess their satisfaction with Iberogast on 5 point Likert scale as "very satisfied", "satisfied", "neither satisfied nor unsatisfied", "unsatisfied", and "very unsatisfied.

SECONDARY OUTCOMES:
Descriptive analyses of demographic data. | At baseline
  Age and sex.
Percentage of patients consulted physician for examination to clarify gastrointestinal complaints. | At baseline
  Functional dyspepsia (FD) and irritable bowel syndrome (IBS) or both.

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.